CLINICAL TRIAL: NCT03529500
Title: Chronic Malnutrition and Oral Health Status in Children Aged One to Five Years
Status: Completed | Type: Observational
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Sandra Kalil Bussadori, Clinical Professor, University of Nove de Julho
Other Study IDs: Malnutrition and oral health
Record Dates: First submitted 2018-04-15; First posted 2018-05-18 (Actual); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: Malnutrition, Child
Keywords: dental caries; saliva; child
MeSH Terms: conditions — Child Nutrition Disorders; Dental Caries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — saliva
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Adequate nutritional status: Dental caries experience was recorded using the dmft index. Active visible white spots were also recorded. Samples of non-stimulated saliva were collected from the participants for five minutes. The salivary flow volume was calculated and expressed as ml/min. After the measurement of salivary flow, an aliquot of 1 ml was transferred to a test tube with 3 ml of hydrochloric acid (HCl 5 mM) for titration and the determination of salivary buffering capacity (SBC).
  Interventions: Diagnostic Test: Caries detection - dmtf index; Diagnostic Test: Saliva flow rate; Diagnostic Test: Saliva Buffering Capacity
- Mild malnutrition: Dental caries experience was recorded using the dmft index. Active visible white spots were also recorded. Samples of non-stimulated saliva were collected from the participants for five minutes. The salivary flow volume was calculated and expressed as ml/min. After the measurement of salivary flow, an aliquot of 1 ml was transferred to a test tube with 3 ml of hydrochloric acid (HCl 5 mM) for titration and the determination of salivary buffering capacity (SBC).
  Interventions: Diagnostic Test: Caries detection - dmtf index; Diagnostic Test: Saliva flow rate; Diagnostic Test: Saliva Buffering Capacity
- Moderate malnutrition: Dental caries experience was recorded using the dmft index. Active visible white spots were also recorded. Samples of non-stimulated saliva were collected from the participants for five minutes. The salivary flow volume was calculated and expressed as ml/min. After the measurement of salivary flow, an aliquot of 1 ml was transferred to a test tube with 3 ml of hydrochloric acid (HCl 5 mM) for titration and the determination of salivary buffering capacity (SBC).
  Interventions: Diagnostic Test: Caries detection - dmtf index; Diagnostic Test: Saliva flow rate; Diagnostic Test: Saliva Buffering Capacity
- Severe malnutrition: Dental caries experience was recorded using the dmft index. Active visible white spots were also recorded. Samples of non-stimulated saliva were collected from the participants for five minutes. The salivary flow volume was calculated and expressed as ml/min. After the measurement of salivary flow, an aliquot of 1 ml was transferred to a test tube with 3 ml of hydrochloric acid (HCl 5 mM) for titration and the determination of salivary buffering capacity (SBC).
  Interventions: Diagnostic Test: Caries detection - dmtf index; Diagnostic Test: Saliva flow rate; Diagnostic Test: Saliva Buffering Capacity

INTERVENTIONS:
Diagnostic Test: Caries detection - dmtf index — Dental caries experience was recorded using the dmft index, which was employed following the recommendations of the WHO to establish the prevalence and severity of caries. Active visible white spots were also recorded. The examinations were performed in duplicate for each child with the aim of establishing inter-examiner agreement using the Kappa statistic which demonstrated good agreement (K = 0.81).
  The criteria adopted for the determination of prevalence followed by guidelines of the Oral Health Surveys - Basic Methods, 4th edition (WHO, 1997) described in the examiner's manual and annotator's manual produced by the coordination team of the Brazil Oral Health Project. The severity and prevalence of dental caries were determined based on the dmft index.
Diagnostic Test: Saliva flow rate — Samples of non-stimulated saliva were collected from the participants for five minutes using two aspirator tubes connected to a 15-ml Falcon tube. One aspirator tube was positioned under the child's tongue and the other was attached to the aspirator device. After five minutes, the amount of saliva was measured for the determination of salivary flow. Collections were performed between 9 and 11 am and the time of the last meal was recorded. At least a one-hour interval was required between the last meal and the collection of the saliva sample. The volume of saliva was measured. The salivary flow volume was calculated and expressed as ml/min. The following categories were considered in the analysis of salivary flow: < 0.1 ml/min = xerostomia; 0.1 to 0.6 ml/min = very low flow; 0.7 to 0.9 mL/min low flow; 1.0 to 2.0 ml/min = normal flow; and > 2.0 ml/min = high flow.
Diagnostic Test: Saliva Buffering Capacity — an aliquot of 1 ml was transferred to a test tube with 3 ml of hydrochloric acid (HCl 5 mM) for titration and the determination of salivary buffering capacity (SBC). The saliva/acid solution was shaken in a q 220 vortex tube agitator (Quimis, Diadema, SP, Brazil) for 15 seconds. Next, pH was determined in a portable pH meter (KASVI K39-0014P, Curitiba, PR, Brazil) for the determination of the SBC. The following categories were considered: ≥ 5.5 = very good buffering capacity; 5.4 to 5.0 = good buffering capacity; 4.9 to 4.5 = medium good buffering capacity; 4.4 to 4.0 = low buffering capacity; and ≤ 3.9 very low buffering capacity.

SUMMARY:
Malnutrition is a public health problem that can exert a negative impact on the general and oral health of children. The aim of the present study was to evaluate the effect of chronic malnutrition on the oral health of children aged one to five years. An observational, analytical, cross-sectional study was conducted at the Nutritional Recovery Center and involved 82 children between 12 and 71 months of age. Nutritional status was evaluated using anthropometric indicators and oral health status was measured using the dmft index. Non-stimulated saliva was collected. Flow rate and buffering capacity was then measured with the aid of a pH meter.

DETAILED DESCRIPTION:
Malnutrition is a public health problem that can exert a negative impact on the general and oral health of children. The aim of the present study was to evaluate the effect of chronic malnutrition on the oral health of children aged one to five years. An observational, analytical, cross-sectional study was conducted at the Nutritional Recovery Center and involved 82 children between 12 and 71 months of age. Nutritional status was evaluated using anthropometric indicators. The children were weighed on a previously calibrated electronic scale (capacity: 150 kg; precision: 100 g) barefoot and wearing light clothing in the presence of the mother or caregiver. Height was determined using a non-flexible metric tape (maximum length: 2 m; precision: 0.1 cm). Each measurement was made twice and the mean was used for the calculation height for age, weight for height and weight for age. The guidelines of the World Health Organization, were the reference for the evaluation of nutritional status. Oral health status was measured using the dmft index. The criteria adopted for the determination of prevalence followed by guidelines of the Oral Health Surveys - Basic Methods, 4th edition - described in the examiner's manual and annotator's manual produced by the coordination team of the Brazil Oral Health Project. Non-stimulated saliva was collected and Flow rate and buffering capacity was then measured with the aid of a pH meter. The salivary flow volume was calculated and expressed as ml/min. The following categories were considered in the analysis of salivary flow: < 0.1 ml/min = xerostomia; 0.1 to 0.6 ml/min = very low flow; 0.7 to 0.9 mL/min low flow; 1.0 to 2.0 ml/min = normal flow; and > 2.0 ml/min = high flow. The following categories were considered: ≥ 5.5 = very good buffering capacity; 5.4 to 5.0 = good buffering capacity; 4.9 to 4.5 = medium good buffering capacity; 4.4 to 4.0 = low buffering capacity; and ≤ 3.9 very low buffering capacity.

ELIGIBILITY:
Inclusion Criteria:

Children aged one to five years enrolled at the Center for Educational and Nutrition Recovery.

Statement of informed consent signed by parents/guardians. Clinical diagnosis of malnutrition.

Exclusion Criteria:

Children aged one to five years not enrolled at the Center for Educational and Nutrition Recovery.

Children whose Parents/guardians did not sign a statement of informed consent.

Ages: 12 Months to 71 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: This cross-sectional study will use a sample of children aged 12 to 71 months of the 7th Administrative Region of Maceió. This region is one of the poorest region in Maceió. The children's parents/guardians will be interviewed at the Center for Educational and Nutrition Recovery (CREN) in the city of Maceió, state of Alagoas, Brazil. The sample size was estimated considering a prevalence of malnutrition of about 20% in children under 6 years old, with statistical power of 80% and 95% significance, resulting in a sample of 100 children.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2017-02-02 (Actual); Primary Completion 2017-04-27 (Actual); Study Completion 2017-07-27 (Actual)

PRIMARY OUTCOMES:
Weight Measurement | 4 weeks
  The children were weighed on a previously calibrated electronic scale (capacity: 150 kg; precision: 100 g) barefoot and wearing light clothing in the presence of the mother or caregiver.
Height Measurement | 4 weeks
  Height was determined using a non-flexible metric tape (maximum length: 2 m; precision: 0.1 cm).

SECONDARY OUTCOMES:
Evaluation of dental caries | 2 weeks
  Dental Caries - dental caries experience was recorded using the dmft index, which was employed following the recommendations of the WHO (WHO, 2007) to establish the prevalence and severity of caries.
Evaluation of saliva flow rate | 4 weeks
  saliva flow rate - The salivary flow volume was calculated and expressed as ml/min. The following categories were considered in the analysis of salivary flow: < 0.1 ml/min = xerostomia; 0.1 to 0.6 ml/min = very low flow; 0.7 to 0.9 mL/min low flow; 1.0 to 2.0 ml/min = normal flow; and > 2.0 ml/min = high flow.
Evaluation of saliva buffering capacity | 4 weeks
  salivary buffering capacity - an aliquot of 1 ml was transferred to a test tube with 3 ml of hydrochloric acid (HCl 5 mM) for titration and the determination of salivary buffering capacity (SBC). The saliva/acid solution was shaken in a q 220 vortex tube agitator (Quimis, Diadema, SP, Brazil) for 15 seconds. Next, pH was determined in a portable pH meter (KASVI K39-0014P, Curitiba, PR, Brazil) for the determination of the SBC. The following categories were considered: ≥ 5.5 = very good buffering capacity; 5.4 to 5.0 = good buffering capacity; 4.9 to 4.5 = medium good buffering capacity; 4.4 to 4.0 = low buffering capacity; and ≤ 3.9 very low buffering capacity .

CONTACTS AND LOCATIONS:
Locations (1):
- Nutritional Recovery Center, Maceió, Alagoas, Brazil

IPD SHARING:
Plan to Share IPD: Yes
All IPD will be available after publication of results.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After results publication.
Access Criteria: Depends on the journal criteria

REFERENCES:
- [Background] Black RE, Allen LH, Bhutta ZA, Caulfield LE, de Onis M, Ezzati M, Mathers C, Rivera J; Maternal and Child Undernutrition Study Group. Maternal and child undernutrition: global and regional exposures and health consequences. Lancet. 2008 Jan 19;371(9608):243-60. doi: 10.1016/S0140-6736(07)61690-0. No abstract available. PMID 18207566
- [Background] Folayan MO, Kolawole KA, Oziegbe EO, Oyedele T, Oshomoji OV, Chukwumah NM, Onyejaka N. Prevalence, and early childhood caries risk indicators in preschool children in suburban Nigeria. BMC Oral Health. 2015 Jun 30;15:72. doi: 10.1186/s12903-015-0058-y. PMID 26123713
- [Background] Hallett KB, O'Rourke PK. Pattern and severity of early childhood caries. Community Dent Oral Epidemiol. 2006 Feb;34(1):25-35. doi: 10.1111/j.1600-0528.2006.00246.x. PMID 16423028
- [Background] Jamelli SR, Rodrigues CS, de Lira PI. Nutritional status and prevalence of dental caries among 12-year-old children at public schools: a case-control study. Oral Health Prev Dent. 2010;8(1):77-84. PMID 20480058
- [Background] Oliveira LB, Sheiham A, Bonecker M. Exploring the association of dental caries with social factors and nutritional status in Brazilian preschool children. Eur J Oral Sci. 2008 Feb;116(1):37-43. doi: 10.1111/j.1600-0722.2007.00507.x. PMID 18186730
- [Background] Palmer CA, Kent R Jr, Loo CY, Hughes CV, Stutius E, Pradhan N, Dahlan M, Kanasi E, Arevalo Vasquez SS, Tanner AC. Diet and caries-associated bacteria in severe early childhood caries. J Dent Res. 2010 Nov;89(11):1224-9. doi: 10.1177/0022034510376543. Epub 2010 Sep 21. PMID 20858780
- [Background] Ramos CV, Dumith SC, Cesar JA. Prevalence and factors associated with stunting and excess weight in children aged 0-5 years from the Brazilian semi-arid region. J Pediatr (Rio J). 2015 Mar-Apr;91(2):175-82. doi: 10.1016/j.jped.2014.07.005. Epub 2014 Nov 6. PMID 25449789
- [Background] Torres SR, Nucci M, Milanos E, Pereira RP, Massaud A, Munhoz T. Variations of salivary flow rates in Brazilian school children. Braz Oral Res. 2006 Jan-Mar;20(1):8-12. doi: 10.1590/s1806-83242006000100003. Epub 2006 May 22. PMID 16729168
- [Result] Bissar A, Schiller P, Wolff A, Niekusch U, Schulte AG. Factors contributing to severe early childhood caries in south-west Germany. Clin Oral Investig. 2014;18(5):1411-8. doi: 10.1007/s00784-013-1116-y. Epub 2013 Oct 11. PMID 24114252
- [Result] Brouwer F, Askar H, Paris S, Schwendicke F. Detecting Secondary Caries Lesions: A Systematic Review and Meta-analysis. J Dent Res. 2016 Feb;95(2):143-51. doi: 10.1177/0022034515611041. Epub 2015 Oct 13. PMID 26464398
- [Result] Correa-Faria P, Martins-Junior PA, Vieira-Andrade RG, Marques LS, Ramos-Jorge ML. Factors associated with the development of early childhood caries among Brazilian preschoolers. Braz Oral Res. 2013 Jul-Aug;27(4):356-62. doi: 10.1590/S1806-83242013005000021. PMID 23780495
- [Result] Das D, Misra J, Mitra M, Bhattacharya B, Bagchi A. Prevalence of dental caries and treatment needs in children in coastal areas of West Bengal. Contemp Clin Dent. 2013 Oct;4(4):482-7. doi: 10.4103/0976-237X.123048. PMID 24403793
- [Result] Fontana M. The Clinical, Environmental, and Behavioral Factors That Foster Early Childhood Caries: Evidence for Caries Risk Assessment. Pediatr Dent. 2015 May-Jun;37(3):217-25. PMID 26063551
- [Result] Johansson I, Lenander-Lumikari M, Saellstrom AK. Saliva composition in Indian children with chronic protein-energy malnutrition. J Dent Res. 1994 Jan;73(1):11-9. doi: 10.1177/00220345940730010101. PMID 8294612
- [Result] Moynihan P, Petersen PE. Diet, nutrition and the prevention of dental diseases. Public Health Nutr. 2004 Feb;7(1A):201-26. doi: 10.1079/phn2003589. PMID 14972061
- [Result] Psoter WJ, Reid BC, Katz RV. Malnutrition and dental caries: a review of the literature. Caries Res. 2005 Nov-Dec;39(6):441-7. doi: 10.1159/000088178. PMID 16251787
- [Result] Psoter WJ, Spielman AL, Gebrian B, St Jean R, Katz RV. Effect of childhood malnutrition on salivary flow and pH. Arch Oral Biol. 2008 Mar;53(3):231-7. doi: 10.1016/j.archoralbio.2007.09.007. Epub 2007 Nov 5. PMID 17983611
- [Result] Samnieng P, Ueno M, Shinada K, Zaitsu T, Wright FA, Kawaguchi Y. Association of hyposalivation with oral function, nutrition and oral health in community-dwelling elderly Thai. Community Dent Health. 2012 Mar;29(1):117-23. PMID 22482262
- [Result] Sheetal A, Hiremath VK, Patil AG, Sajjansetty S, Kumar SR. Malnutrition and its oral outcome - a review. J Clin Diagn Res. 2013 Jan;7(1):178-80. doi: 10.7860/JCDR/2012/5104.2702. Epub 2013 Jan 1. PMID 23449967